CLINICAL TRIAL: NCT03515824
Title: A Phase 1 Study of MK-1697 in Participants With Advanced Solid Tumors
Brief Title: Study of MK-1697 in Participants With Advanced Solid Tumors (MK-1697-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1697-001; MK1697-001 (Other: Merck)
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); PD-1; PDL1; PD-L1
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: MK-1696 20 mg (Experimental): Participants received 20 mg of MK-1697 by intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-1697
- Part A: MK-1697 65 mg (Experimental): Participants received 65 mg of MK-1697 by IV infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-1697
- Part A: MK-1697 200 mg (Experimental): Participants received 200 mg of MK-1697 by IV infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-1697
- Part B: Expansion Cohort (Experimental): Participants with select tumor types were to receive MK-1697 at the RP2D by IV infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-1697

INTERVENTIONS:
Biological: MK-1697 — Administered by IV infusion on Day 1 of each 21-day cycle

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of MK-1697. There are 2 parts in this study: dose escalation to determine the recommended phase 2 dose (RP2D) and confirm the RP2D (Part A) and cohort expansion to determine preliminary efficacy in participants with colorectal cancer (CRC) or head and neck squamous cell cancer (HNSCC) (Part B). No formal hypothesis testing will be done in this study.

ELIGIBILITY:
Inclusion Criteria:

* For Part A; has a histologically- or cytologically-confirmed advanced/metastatic solid tumor and has received, been intolerant to, or been ineligible for all treatments known to confer clinical benefit
* For Part B: has 1 of the following histologically or cytologically confirmed tumor types that are anti-programmed cell death protein 1 (anti PD-1)/anti-programmed death-ligand 1 (anti PD-L1) treatment naive:

  * CRC originating in either the colon or rectum that is locally advanced unresectable or metastatic (ie, Stage IV) and that has received, and progressed on, all available standard-of-care therapies including fluoropyrimidine, oxaliplatin, and irinotecan
  * HNSCC that is considered incurable by local therapies. The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx. Participants may not have a primary tumor site of nasopharynx (any histology). Also, participants must have progressed after receiving platinum-containing systemic therapy
* Has measurable disease by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
* Has an evaluable baseline tumor sample (either a recent or archival) for analysis
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has central venous access (eg, portacath, Hickman line, or peripherally inserted central catheter [PICC] line) currently inserted or be considered medically fit for and willing to undergo the insertion of such a device
* Is not pregnant or breastfeeding
* Female participants of childbearing potential must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period

Exclusion Criteria:

* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years with the exception of participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer, or other in-situ cancers
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction to treatment with any monoclonal antibody and/or components of the study treatment
* Has an active infection requiring therapy
* Has a history of interstitial lung disease
* Has a history of (noninfectious) pneumonitis that required steroids or current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has known human immunodeficiency virus (HIV) and/or Hepatitis B or C infections, or known to be positive for Hepatitis B antigen/Hepatitis B virus deoxyribonucleic acid (DNA) or Hepatitis C Antibody or ribonucleic acid (RNA)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with participation, make administration of the study treatments hazardous, or make it difficult to monitor adverse effects in the opinion of the treating investigator
* Has a history or current evidence of severe cardiovascular disease, ie, arrhythmias requiring chronic treatment, congestive heart failure (New York Heart Association [NYHA] Class III or IV) or symptomatic ischemic heart disease.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has not fully recovered from any effects of major surgery without significant detectable infection. Surgeries that required general anesthesia must be completed at least 2 weeks before first study treatment administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study treatment administration and participants should be recovered
* Has known microsatellite instability (MSI) high or mismatch repair genes (MMR) deficient colorectal cancer. If a participant's MSI status is unknown, a paired blood sample for MSI in addition to biomarker testing is required to determine MSI status retrospectively (for the CRC expansion cohort only)
* Has a positive pregnancy test within 72 hours before the first dose of study treatment
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study therapy, or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any adverse events that were due to cancer therapeutics administered more than 4 weeks earlier
* Has received prior therapy with an anti-Lymphocyte-activation gene 3 (LAG-3) agent
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Has undergone a prior stem cell or bone marrow transplant within the last 5 years
* Is expected to require any other form of antineoplastic therapy while on study
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Scientia Clinical Research ( Site 0100), Randwick, New South Wales, Australia
- Queen Mary Hospital ( Site 0200), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 22 participants allocated received study treatment (All Treated Population) and were evaluable for all safety analysis. Expansion Cohort (Part B) did not enroll any participants.
Groups:
- Part A: MK-1697 20 mg: Participants received 20 mg of MK-1697 by IV infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years).
- Part B: Expansion Cohort: Participants with select tumor types were to receive MK-1697 at the RP2D by IV infusion on Day 1 of each 21-day cycle for up to 35 administrations (up to approximately 2 years). No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg | Part B: Expansion Cohort
Started | 3 | 4 | 15 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 15 | 0
Not completed — Death | 3 | 2 | 6 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 6 | 0
Not completed — Status not recorded | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Part B since study was terminated at the completion of Part A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg | Total
Number analyzed (Participants) | 3 | 4 | 15 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (8.4) | 57.3 (19.8) | 51.8 (14.5) | 54.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 10 | 12
  Male | 2 | 3 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 15 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 9 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Dose Limiting Toxicity (DLT) During Cycle 1
Description: The following toxicities were considered a DLT, if assessed as related to study treatment: Grade (Gr) 4 non-hematologic toxicity (T); Gr 4 hematologic T for ≥7 days; Gr 4 thrombocytopenia; Gr 3 thrombocytopenia with bleeding; ≥Gr 3 non-hematologic clinical AE except fatigue for ≤3 days, Gr 3 nausea, vomiting, or diarrhea for >72 hours despite anti-emetics/diarrheals, or other supportive care; Gr 3 rash without corticosteroids/anti-inflammatory agents use per standard of care; Gr 3/4 non-hematologic laboratory value if: medical intervention is required, abnormality leads to hospitalization, persists for >1 week, or abnormality results in drug-induced liver injury; Gr 3 or 4 febrile neutropenia; treatment-related T causing discontinuation; inability to administer ≥75% of planned dose due to drug-related tolerability; Gr 5 T; delay in Cycle 2 start by >2 weeks due to T. Pool-adjacent violators algorithm was used to estimate DLT rate & Bayesian method for 80% confidence intervals (CIs).
Time Frame: Up to 21 days of Cycle 1 (cycle length = 21 days)
Population: All Part A participants who received at least 1 dose of study treatment and finished Cycle 1 without a DLT or experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 3 | 13
Participants | 0 | 0 | 2
Statistical Analysis 1: Comparison: Part A: MK-1697 20 mg; Test type: Other — Bayesian posterior credible interval; Pooled-adjacent-violator algorithm = 0.0, 80% CI 2-sided [0.0 to 33.1]
Statistical Analysis 2: Comparison: Part A: MK-1697 65 mg; Test type: Other — Bayesian posterior credible interval; Pooled-adjacent-violator algorithm = 0.0, 80% CI 2-sided [0.0 to 33.1]
Statistical Analysis 3: Comparison: Part A: MK-1697 200 mg; Test type: Other — Bayesian posterior credible interval; Pooled-adjacent-violator algorithm = 15.4, 80% CI 2-sided [5.8 to 30.2]

2. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experienced at least one AE were presented.
Time Frame: Up to approximately 9 months
Population: All Part A participants who received at least one dose of study treatment. Expansion Cohort (Part B) did not enroll any participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
Participants | 3 | 4 | 14

3. Primary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinued study intervention due to an AE were presented.
Time Frame: Up to approximately 8 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
Participants | 0 | 1 | 3

4. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
Description: An objective response was defined as a complete response (CR: Disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by the investigator based on RECIST 1.1 following administration of MK-1697. ORR was reported as percentage of participants who experienced an CR or PR after administration of MK-1967. The exact method based on the binomial distribution (Clopper-Pearson interval) was used to estimate ORR and its associated 95%CIs.
Time Frame: Up to approximately 18 months (through End of Trial data cut-off 18 Feb 2020)
Population: All Part A participants with a baseline scan that demonstrated measurable disease by the investigator's assessment, and who received at least 1 dose of study treatment were evaluated. Expansion Cohort (Part B) did not enroll any participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
Percentage of Participants | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Part A: MK-1697 20 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate (ORR) = 0.0, 95% CI 2-sided [0.0 to 70.8]
Statistical Analysis 2: Comparison: Part A: MK-1697 65 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate (ORR) = 0.0, 95% CI 2-sided [0.0 to 60.2]
Statistical Analysis 3: Comparison: Part A: MK-1697 200 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate (ORR) = 0.0, 95% CI 2-sided [0.0 to 21.8]

5. Secondary Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria In Solid Tumors Version 1.1 for Immune-based Therapeutics (iRECIST)
Description: An objective response was defined as an immune-based complete response (iCR: Disappearance of all target lesions) or immune-based partial response (iPR: At least a 30% decrease in the sum of diameters of target lesions). ORR was reported as percentage of participants who experienced an iCR or iPR after administration of MK-1967. Participants were initially assessed for progressive disease (PD : ≥20% increase in sum of diameters [SD] of target lesions or relative increase of 20%, sum must demonstrate an absolute increase of ≥5 mm or appearance of one/more new lesions) per RECIST 1.1 by local site investigator; later verified by central imaging vendor. Investigator could elect to continue treatment and tumor assessment repeated 4-8 weeks later to confirm PD by iRECIST. The exact method based on the binomial distribution (Clopper-Pearson interval) was used to estimate ORR and its associated 95%CIs.
Time Frame: Up to approximately 18 months (through End of Trial data cut-off 18 Feb 2020)
Population: All Part A participants that demonstrated PD by RECIST 1.1 per investigator's assessment, who received at least 1 dose of study treatment and were complaint with study procedures. Expansion Cohort (Part B) did not enroll any participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 2 | 3 | 11
Percentage of Participants | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Part A: MK-1697 20 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate (ORR) = 0, 95% CI 2-sided [0.0 to 84.2]
Statistical Analysis 2: Comparison: Part A: MK-1697 65 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate (ORR) = 0.0, 95% CI 2-sided [0.0 to 70.8]
Statistical Analysis 3: Comparison: Part A: MK-1697 200 mg; Test type: Other — Clopper Pearson confidence interval method for binomial data; Objective Response Rate )ORR) = 0.0, 95% CI 2-sided [0.0 to 28.5]

6. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC 0-inf) of MK-1697
Description: Serum samples were collected at specified time points for determination of MK-1697 AUC 0-inf. AUC 0-inf was defined as the area under the concentration-time curve of MK-1697 from time zero to infinity for all participants in Part A for each dose group.
Time Frame: Cycle 1-3: Days 1, 2 (only Cycle 1), 3, 8, 15 - predose and postdose at 10 minutes, 2 hours (cycle length = 21 days)
Population: All Part A participants who were compliant with the study procedures and have AUC 0-inf data available from at least one treatment. Participants vary across cycles due to availability of adequate data to allow computation of AUC 0-inf in each cycle based on compliance with study procedures. Expansion Cohort (Part B) did not enroll any participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ng/mL
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
Day*ng/mL
  Cycle 1: number analyzed (Participants) | 3 | 3 | 14
  Cycle 1 | 29500 (106.3) | 143000 (40.9) | 456000 (25.6)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 11
  Cycle 2 | 23400 (65.4) | 168000 (42.1) | 499000 (47.9)
  Cycle 3: number analyzed (Participants) | 2 | 3 | 11
  Cycle 3 | 29300 (64.0) | 188000 (53.0) | 555000 (42.1)

7. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration (AUC 0-last) Measured of MK-1697
Description: Serum samples were collected at specified time points for determination of AUC 0-last of MK-1697. AUC 0-last was defined as the area under the concentration-time curve of MK-1697 from time zero to the last concentration of MK-1697 measured for all participants in Part A for each dose group.
Time Frame: Cycles 1, 2, and 3: predose, 10 minutes and 2 hours post-dose (cycle length = 21 days)
Population: All Part A participants who were compliant with the study procedures and have AUC 0-last data available from at least one treatment. Participants vary across cycles due to availability of adequate data to allow computation of AUC 0-last in each cycle based on compliance with study procedures. Expansion Cohort (Part B) did not enroll any participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ng/mL
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
Day*ng/mL
  Cycle 1 | 27700 (103.0) | 99000 (59.7) | 280000 (143.1)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 11
  Cycle 2 | 28000 (60.9) | 141000 (34.3) | 418000 (38.4)
  Cycle 3: number analyzed (Participants) | 3 | 3 | 11
  Cycle 3 | 8220 (763.8) | 162000 (49.8) | 442000 (35.1)

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of MK-1697
Description: Serum samples were collected at specified time points for determination of MK-1697 Cmax. Cmax was defined as the maximum concentration of MK-1697 reached for all participants in Part A for each dose group.
Time Frame: Cycle 1-3: Days 1, 2 (only Cycle 1), 3, 8, 15 - predose and postdose at 10 minutes, 2 hours (cycle length = 21 days)
Population: All Part A participants who were compliant with the study procedures and have Cmax data available from at least one treatment. Participants vary across cycles due to early discontinuation and not completing planned assessments. Expansion Cohort (Part B) did not enroll any participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
ng/mL
  Cycle 1 | 5520 (89.9) | 16900 (31.2) | 60200 (12.5)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 11
  Cycle 2 | 5850 (37.5) | 21800 (31.5) | 58500 (27.8)
  Cycle 3: number analyzed (Participants) | 3 | 3 | 11
  Cycle 3 | 5560 (41.4) | 22500 (33.9) | 61200 (18.7)

9. Secondary Outcome: Minimum Serum Concentration (Cmin) of MK-1697
Description: Serum samples were collected pre-dose at specified time points (Cycles 1, 2, 3, 5, 7, and 11) for the determination of MK-1697 Ctrough (may also be referred to as Cmin) per protocol. Ctrough was defined as the lowest concentration of MK-1697 reached before the next dose was administered. Serum Ctrough of MK-1697 was reported for all participants in Part A for each dose group.
Time Frame: Cycles 1-3, 5, 7, 11: Days 1, 2 (only Cycle 1), 3, 8, 15 - predose and postdose at 10 minutes, 2 hours (cycle length = 21 days)
Population: All Part A participants who were compliant with the study procedures and have Cmin data available from at least one treatment. Participants vary across cycles due to early discontinuation and not completing planned assessments. Expansion Cohort (Part B) did not enroll any participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
Number analyzed (Participants) | 3 | 4 | 15
ng/mL
  Cycle 1: number analyzed (Participants) | 3 | 4 | 10
  Cycle 1 | 127 (995.6) | 1310 (107.0) | 3230 (870.7)
  Cycle 2 | 125 (556.0) | 2210 (59.6) | 5350 (190.0)
  Cycle 3: number analyzed (Participants) | 1 | 4 | 9
  Cycle 3 | 566 (NA) — %GCV could not be calculated when n<2 | 2390 (61.8) | 7000 (82.0)
  Cycle 5: number analyzed (Participants) | 1 | 2 | 3
  Cycle 5 | 544 (NA) — %GCV could not be calculated when n<2 | 2540 (129.0) | 9590 (43.4)
  Cycle 7: number analyzed (Participants) | 1 | 2 | 0
  Cycle 7 | 580 (NA) — %GCV could not be calculated when n<2 | 3000 (79.4) |
  Cycle 11: number analyzed (Participants) | 1 | 0 | 0
  Cycle 11 | 631 (NA) — %GCV could not be calculated when n<2 |  |

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected for up to approximately 9 months. All-cause mortality and serious AEs were collected for up to approximately 14 months.
Description: All-Cause Mortality reported for all enrolled participants. Serious AEs and Other AEs were reported for all enrolled participants who received at least 1 dose of study treatment. No participants were enrolled in Part B since study was terminated at the completion of Part A.
Arm/Group | Part A: MK-1697 20 mg | Part A: MK-1697 65 mg | Part A: MK-1697 200 mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/4 | 6/15
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 7/15
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MK-1697 20 mg (N=3) | Part A: MK-1697 65 mg (N=4) | Part A: MK-1697 200 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MK-1697 20 mg (N=3) | Part A: MK-1697 65 mg (N=4) | Part A: MK-1697 200 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 4 (7)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (3) | 2 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT03515824/Prot_SAP_000.pdf